CLINICAL TRIAL: NCT02999035
Title: Validation of a Newly Developed Liquid Jet Aesthesiometer
Status: Completed | Type: Observational
Sponsor: University of Applied Sciences and Arts Northwestern Switzerland (Other)
Responsible Party: Principal Investigator, Remo Poffa, Study coordinator, University of Applied Sciences and Arts Northwestern Switzerland
Other Study IDs: 2016-01867
Record Dates: First submitted 2016-12-14; First posted 2016-12-21 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Ocular Surface Disease
Keywords: ocular surface sensitivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- corneal sensitivity measurement: Air jet aesthesiometry and liquid jet aesthesiometry:
  All patients will receive the same intervention of corneal sensitivity measurement with air jet aesthesiometry and liquid jet aesthesiometry.
  Thresholds represent the intensity of air / liquid jet that can just be perceived by the patients.

SUMMARY:
A new liquid jet aesthesiometer prototype was developed with the aim to measure ocular surface sensitivity by employing a liquid jet.

This study aims to validate this new prototype by means of correlating its measurement with a previously validated air jet aesthesiometer, the non-contact aesthesiometer (NCCA; by Murphy et al. 1996) and by exploring the repeatability of ocular surface sensitivity measurement.

DETAILED DESCRIPTION:
Currently, no aesthesiometer is available that delivers reliable and repeatable measurement of ocular surface sensitivity in a routine clinical setup. The only commercially available Cochet- Bonnet aesthesiometer uses a tactile-mechanical stimulus (the tip of a nylon thread), which can cause a microerosion when applied to the corneal surface. Additional disadvantages represent poor stimulus reproducibility, a limited stimulus bandwidth and the influence of humidity and age on the bending capibility of the nylon thread. For research purposes prototypes of non-contact air aesthesiometers (eg by Murphy et al. and Belmonte et al) are being used.

This study aims to correlate ocular surface sensitivity measurements of a newly developed prototype, the liquid jet aesthesiometer, with the non-contact air jet aesthesiometer by Murphy et al. 1996 and to explore its repeatability of measurement.

In this repeated measures design 60 subjects participate in corneal sensitivity measurements during two appointments with each described aesthesiometer.

ELIGIBILITY:
Inclusion Criteria:

* Ocular surface index score < 13.0

Exclusion Criteria:

* systemic disease such as diabetes, diseases, injuries and operations in the anterior segment of the eye
* systemic medication and / or eyedrops / ointments that may have an influence of the tearfilm.
* contact lens wear less than 48 hours before commencement of study measurements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 healthy subjects within age range of 18-30 years 30 healthy subjects within age range of 50-65 years
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Correlation with air jet aesthesiometry | two measurements / repeated measures within one month
  correlation between corneal sensitivity measurements between liquid jet and air jet aesthesiometry

SECONDARY OUTCOMES:
repeatability of corneal sensitivity measurement with new prototype | two measurements / repeated measures within one month
  repeatability of corneal sensitivity measurement with liquid jet aesthesiometry

CONTACTS AND LOCATIONS:
Overall Officials: Remo Poffa, MSc., Principal Investigator — University of Applied Sciences and Arts Northwestern Switzerland

IPD SHARING:
Plan to Share IPD: No
individual participant data will not be made available to other researchers. The statistical analysis of the data overall will be however published, but individual participant data will not be discussed.

REFERENCES:
- [Background] Murphy PJ, Patel S, Marshall J. A new non-contact corneal aesthesiometer (NCCA). Ophthalmic Physiol Opt. 1996 Mar;16(2):101-7. PMID 8762770
- [Background] COCHET P, BONNET R. [Corneal esthesiometry. Performance and practical importance]. Bull Soc Ophtalmol Fr. 1961 Jul-Aug;6:541-50. No abstract available. French. PMID 13880071
- [Background] Belmonte C, Acosta MC, Schmelz M, Gallar J. Measurement of corneal sensitivity to mechanical and chemical stimulation with a CO2 esthesiometer. Invest Ophthalmol Vis Sci. 1999 Feb;40(2):513-9. PMID 9950612